CLINICAL TRIAL: NCT05568303
Title: The Effect of Cognitive Behavioral Therapy on Psychological Distress Among Mothers of Children With Autism Spectrum Disorders: The Role of Problem-Solving Appraisal
Brief Title: the Role of Problem Solving in Cognitive Behavioral Therapy for Mothers With Autistic Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jouf University (Other)
Responsible Party: Principal Investigator, Enas Mahrous AbdelAziz, assistant professor, Jouf University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 62
Record Dates: First submitted 2022-10-01; First posted 2022-10-05 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Cognitive Behavioral Therapy and Problem Solving; Autism Disorders and Maternal Stress
Keywords: Autism disorders, maternal stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study ( interventional ) group (Experimental): this group received 8 sessions of CBT
  Interventions: Behavioral: CBT techniques
- Control group (No Intervention): they will receive on intervention sessions or any education researchers makes meeting every month to answer any questions and to maintain continuity of relation with participants

INTERVENTIONS:
Behavioral: CBT techniques — through CBT sessions , the participants apply problem solving process in managing their stressors . examining the role of cognitions, emotions, and behaviors to form cause and effect relationship of participants psychological distress
  Arms: study ( interventional ) group

SUMMARY:
Cognitive behavioral therapy sessions can effectively reduce distress in mothers of children with autism. here we emphasize on the role of problem solving appraisal in CBT sessions to improve problem solving skills ability and minimize psychological distress . pre- intervention assessment (T1) for all participants , then designed 8 sessions for study group will apply .

post intervention assessment (T2) will conduct immediately after CBT sessions

DETAILED DESCRIPTION:
mothers of children with autistic spectrum disorders have a lots of burdens due to child symptoms its, lack of availability of services and limited resources , thus in turn lead them to become unable to face problems/stressors and to be psychological distress. CBT is an effective therapy to minimize stress, anxiety and depression. Mothers who participated in the study recruited from three governmental hospitals that has an out patients clinics specialized in autism and other developmental disorders for children at ElBehairah governate , Egypt . Based on inclusion and exclusion criteria for mothers and their children, mothers informed about the nature of the study and their benefits for participations. assessment tools will use ; depression ,anxiety and stress scale (DAS) and problem solving inventory (PSI). First assessment will occur , then randomly the participants divide into either study ( intervention) group or control group .CBT sessions will provide for study group to enhance their problem solving ability and psychological state. Second assessment (T2) will occur after finishing program sessions for all participants

ELIGIBILITY:
Inclusion Criteria:

Mothers caregivers who have:

* A child with autism spectrum disorders diagnosed science at least 6 months , and her/ his diagnosis done by a psychiatrist
* Just one child with autistic disorder
* Their ages between 20-50 years old
* Did not expose to previous interventional / rehabilitation programs for his/her child.

Exclusion Criteria for mothers:

* have a diagnosis of any of psychiatric disorders
* Being absent more than three sessions in study group

Exclusion criteria for children: if they have:

* Intelligence level below 70
* Have severe deterioration
* Receive psychiatric medication
* Have multiple disorders

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — only mothers of autistics children's involve
Enrollment: 60 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Change in mean scores of psychological distress scores among study group post intervention | two months
  Change in mean scores of psychological distress
Change in mean scores of problem solving skills inventor among study group post intervention | 2 months
  Change in mean scores of problem solving skills inventory

CONTACTS AND LOCATIONS:
Overall Officials: Enas M Abdelaziz, PhD, Principal Investigator — Jouf University
Locations (2):
- Governmental Clinic, Behera Governate, Beera, Egypt
- Enas Mahrous Abdelaziz, JOUF, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
based on request from principle investigator